CLINICAL TRIAL: NCT04161001
Title: A Multi-center, Randomized, Double-Blind, Phase III Clinical Trial to Evaluate the Efficacy and Safety of DWJ1451 in Patients With Hypertension and Dyslipidemia
Brief Title: Clinical Trail to Evaluate the Efficacy and Safety of DWJ1451
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW_DWJ1451301
Record Dates: First submitted 2019-11-07; First posted 2019-11-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Hypertension, Dyslipidemia
MeSH Terms: conditions — Hypertension; Dyslipidemias | interventions — Amlodipine; olmesartan; Drug Combinations; Ezetimibe; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Amlodpine, Olmesartan, Rosuvastatin, Ezetimibe (Experimental): co-administration of Olmesartan, Amlodipine and Rosuvastatin, Ezetimibe
  Interventions: Drug: Amlodipine/Olmesartan 10/40mg (Combination drug), Ezetimibe/Rosuvastatin 10/20mg(Combination drug)
- Olmesartan, Rosuvastatin, Ezetimibe (Placebo Comparator): co-administration of Olmesartan and Rosuvastatin, Ezetimibe
  Interventions: Drug: Olmesartan 40mg, Ezetimibe/Rosuvastatin 10/20mg(Combination drug)
- Amlodpine, Olmesartan (Placebo Comparator): co-administration of Olmesartan, Amlodipine
  Interventions: Drug: Amlodipine/Olmesartan 10/40mg (Combination drug)

INTERVENTIONS:
Drug: Amlodipine/Olmesartan 10/40mg (Combination drug), Ezetimibe/Rosuvastatin 10/20mg(Combination drug) — co-administration of Sevikar tab. 10/40mg(Amlodipine/Olmesartan 10/40mg), Rosuzet Tab. 10/20mg(Ezetimibe/Rosuvastatin 10/20mg) and placebo of Olmetec Tab. 40mg(Olmesartan 40mg)
  Arms: Amlodpine, Olmesartan, Rosuvastatin, Ezetimibe
Drug: Olmesartan 40mg, Ezetimibe/Rosuvastatin 10/20mg(Combination drug) — co-administration of Olmetec tab. 40mg(Olmesartan 40mg), Rosuzet Tab. 10/20mg(Ezetimibe/Rosuvastatin 10/20mg) and placebo of Sevikar tab. 10/40mg (Amlodipine/Olmesartan 10/40mg)
  Arms: Olmesartan, Rosuvastatin, Ezetimibe
Drug: Amlodipine/Olmesartan 10/40mg (Combination drug) — co-administration of Sevikar tab. 10/40mg(Amlodipine/Olmesartan 10/40mg, and placebo of Rosuzet Tab. 10/20mg(Ezetimibe/Rosuvastatin 10/20mg), Olmetec Tab. 40mg(Olmesartan 40mg)
  Arms: Amlodpine, Olmesartan

SUMMARY:
* the change of sitSBP based on baseline between Treatment arm and control 1 arm [ Time Frame: 8 weeks ]
* the change of LDL-C based on baseline between Treatment arm and control2 arm [ Time Frame: 8 weeks ]

ELIGIBILITY:
Inclusion Criteria:

* Age 19 to 80 years
* patients with hypertension and hyperlipidemias

Exclusion Criteria:

* orthostatic hypotension
* History of ventricular tachycardia, atrial fibrillation
* uncontrolled diabetes mellitus

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Estimated)
Dates: Start 2019-11-20 (Estimated); Primary Completion 2021-11-20 (Estimated); Study Completion 2022-02-02 (Estimated)

PRIMARY OUTCOMES:
the change of MSSBP based on baseline between Treatment arm and control 1 arm | 8 weeks
the change of LDL-C based on baseline between Treatment arm and control2 arm | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea